CLINICAL TRIAL: NCT05647629
Title: Development of Low Back Pain After Total Hip Arthroplasty.
Brief Title: Observational Study of the Development of Low Back Pain After Total Hip Arthroplasty.
Status: Recruiting | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Francisco José Gallego Peñalver, Principal Investigator, Universidad de Zaragoza
Other Study IDs: PI21/346
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain; Hip Osteoarthritis; Arthropathy of Hip
Keywords: Pain; Low back pain; Psoas muscle; Hip arthroplasty
MeSH Terms: conditions — Low Back Pain; Osteoarthritis, Hip; Pain | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total hip arthroplasty — hip prosthesis surgery

SUMMARY:
The investigators are going to observe the appearance of low back pain in patients who have undergone hip prosthesis surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age and under 70 years of age, intervened by CTA due to OAC since January 1, 2010 and before January 1, 2021 and who have developed subsequent lumbar pathology.

Exclusion Criteria (relative/absolute):

* Under 18 years of age at the time of the intervention.
* Over 70 years of age at the time of surgery.
* Previous low back pain.
* Bilateral CTA.
* Previous lower limb or axial fracture.
* Dysmetria.
* Vertebral surgery prior to CTA.
* Scoliosis.
* Scheuermann's disease.
* Neoplasms affecting axial skeleton.
* Bone infections.
* Neurodegenerative disease.
* CTA secondary to fractures.
* CTA replacements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population corresponding to Sector II of Zaragoza, Autonomous Community of Aragon, Spain.
Sampling Method: Probability Sample
Enrollment: 618 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of patients with low back pain | 10 years
  First episode of low back pain

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Francisco José Gallego Peñalver, Valencia
  - Francisco José Gallego Peñalver, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mak D, Chisholm C, Davies AM, Botchu R, James SL. Psoas muscle atrophy following unilateral hip arthroplasty. Skeletal Radiol. 2020 Oct;49(10):1539-1545. doi: 10.1007/s00256-020-03447-3. Epub 2020 May 2. PMID 32361852
- [Background] Morohashi I, Homma Y, Kanda A, Yamamoto Y, Obata H, Mogami A, Obayashi O, Kaneko K. Iliopsoas impingement after revision total hip arthroplasty treated with iliopsoas muscle transection. Ann Med Surg (Lond). 2016 Mar 10;7:30-3. doi: 10.1016/j.amsu.2016.03.004. eCollection 2016 May. PMID 27054031
- [Background] Slater N, Singh R, Senasinghe N, Gore R, Goroszeniuk T, James D. Pressure monitoring of the femoral nerve during total hip replacement: an explanation for iatropathic palsy. J R Coll Surg Edinb. 2000 Aug;45(4):231-3. PMID 11130022
- [Background] Zhu J, Li Y, Chen K, Xiao F, Shen C, Peng J, Chen X. Iliopsoas tendonitis following total hip replacement in highly dysplastic hips: a retrospective study. J Orthop Surg Res. 2019 May 22;14(1):145. doi: 10.1186/s13018-019-1176-z. PMID 31118071
- [Background] Hessmann MH, Hubschle L, Tannast M, Siebenrock KA, Ganz R. [Irritation of the iliopsoas tendon after total hip arthroplasty]. Orthopade. 2007 Aug;36(8):746-51. doi: 10.1007/s00132-007-1094-3. German. PMID 17541541
- [Background] Rasch A, Bystrom AH, Dalen N, Berg HE. Reduced muscle radiological density, cross-sectional area, and strength of major hip and knee muscles in 22 patients with hip osteoarthritis. Acta Orthop. 2007 Aug;78(4):505-10. doi: 10.1080/17453670710014158. PMID 17966005
- [Result] Jorda Llona M, Perez Bocanegra E, Garcia-Mifsud M, Jimeno Bernad R, Ortiz Hernandez R, Castells Ayuso P. [Back school: a simple way to improve pain and postural behaviour]. An Pediatr (Barc). 2014 Aug;81(2):92-8. doi: 10.1016/j.anpedi.2013.11.018. Epub 2013 Dec 28. Spanish. PMID 24380773
- [Derived] Gallego-Penalver FJ, Romero-de-la-Higuera SB, Berdejo Arceiz V, Gomez Trullen EM. Low back pain after total hip arthroplasty: Long-term retrospective cohort study. Rehabilitacion (Madr). 2025 Jul-Sep;59(3):100928. doi: 10.1016/j.rh.2025.100928. Epub 2025 Aug 4. PMID 40763561